CLINICAL TRIAL: NCT04457167
Title: Mastectomy With Retention of the Nipple-areola Complex, Robot-assisted or Not, and / or Immediate or Secondary Reconstruction by Latissimus Dorsi Flap, Robot-assisted or Not.
Brief Title: Mastectomy With Retention of the Nipple-areola Complex, Robot-assisted or Not, and / or Immediate or Seconday Reconstruction by Latissimus Dorsi Flap, Robot-assisted or Not.
Acronym: RMR
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Paoli-Calmettes (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RMR-IPC 2017-039; 2020-A01644-35 (Other: ANSM)
Record Dates: First submitted 2020-06-30; First posted 2020-07-07 (Actual); Last update posted 2020-07-07 (Actual); Status verified 2020-06

CONDITIONS: Mastectomy; Breast Reconstruction
Keywords: robot-assisted; mini-invasive surgery
MeSH Terms: interventions — Robotic Surgical Procedures

STUDY DESIGN:
Intervention Model Description: Phase III, non-randomized, monocentric, observational, prospective trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Robotic surgery (Experimental): Robotic surgery for breast mastectomy with conservation of areolo-nipple plate and immediate or delayed reconstruction by latissimus dorsi flap,
  Interventions: Device: Robot-assisted
- Non robotic surgery (Active Comparator): Non-robotic surgery for breast mastectomy with conservation of areolo-nipple plate and immediate or delayed reconstruction by latissimus dorsi flap,
  Interventions: Procedure: Not robot-assisted surgery

INTERVENTIONS:
Device: Robot-assisted — robot-assisted surgery
  Arms: Robotic surgery
Procedure: Not robot-assisted surgery — Not robot-assisted surgery
  Arms: Non robotic surgery

SUMMARY:
Phase III, non-randomized, monocentric, observational, prospective trial. It is planned to recruit a total of 480 patients, including 240 patients receiving mastectomy with preservation of the nipple-areola complex and 240 patients with a reconstruction with latissimus dorsi flap, or in immediate reconstruction, or during secondary reconstruction.

DETAILED DESCRIPTION:
Phase III, non-randomized, monocentric, observational, prospective trial. It is planned to recruit a total of 480 patients, including 240 patients receiving mastectomy with preservation of the nipple-areola complex and 240 patients with a reconstruction with latissimus dorsi flap, or in immediate reconstruction, or during secondary reconstruction.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old,
2. Signed consent to participate,
3. Women with breast cancer over 18 or at high risk of breast cancer (BRCA 1-2 mutations, PALB2, extensive border lesions)
4. Mastectomy with conservation of the areolo-mammary plaque, or mastectomy without conservation of the areolo-mammary plaque and conservation of the skin case
5. Mastectomy without conservation of the areolo-mammary plate, immediate breast reconstruction by prosthesis,
6. immediate breast reconstruction by autologous latissimus dorsi flap
7. immediate breast reconstruction by latissimus dorsi flap and prosthesis,
8. secondary breast reconstruction by latissimus dorsi flap
9. Affiliation to, or beneficiary of, a social security scheme.

Exclusion Criteria:

1. Patient under 18,
2. Pregnant woman or likely to be (without effective contraception) or breastfeeding,
3. Person in emergency situation, adult person subject to a legal protection measure (adult under guardianship, curatorship or safeguard of justice), or out of state to express his consent,
4. Inability to submit to medical follow-up for the trial for geographic, social or psychological reasons.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 480 (Estimated)
Dates: Start 2020-11-01 (Estimated); Primary Completion 2023-11-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
rate of postoperative early complications | 90 days
  To assess the value of robotic surgery for breast mastectomy with preservation of the nipple-areola complex and immediate or delayed reconstruction by latissimus dorsi flap, with an evaluation of the rate of postoperative early complications (90 postoperative days)

CONTACTS AND LOCATIONS:
Overall Officials: Gilles Houvenaeghel, Principal Investigator — Institut Paoli-Calmettes
Locations (1):
- Institut Paoli-Calmettes, Marseille, France

IPD SHARING:
Plan to Share IPD: No